CLINICAL TRIAL: NCT06110416
Title: Decreasing Post-Operative Nausea and Vomiting in the Bariatric Surgical Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 058.NUR.2020.M
Record Dates: First submitted 2020-11-18; First posted 2023-10-31 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Nausea, Postoperative; Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aromatherapy (Other)
  Interventions: Other: nausea relief inhaler

INTERVENTIONS:
Other: nausea relief inhaler — Aromatherapy and essential oils are an alternative method to controlling post-operative nausea and vomiting after post-surgical intervention.

SUMMARY:
From the research and current studies, post-operative nausea and vomiting is a common complaint after bariatric surgery. Nausea relief inhalers could improve post-operative nausea and vomiting without the need for further medications, subsequently reducing the chance of side effects. This study could help improve patient satisfaction and increase the ability of the patient to ambulate after surgery with the use of a nausea relief inhaler.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting is a very common and uncomfortable issue that occurs after bariatric surgery. 65% of patients have post-operative nausea and vomiting. Compared to previously published results, this percentage was higher than patients undergoing ambulatory surgery. The most common start of post-operative nausea and vomiting was in the first six hours but continued to increase during the first 24 hours. Post-operative nausea and vomiting inhibits early mobilization for the patient affected. Even patients that received nausea and vomiting prophylaxis at the optimal amount had an 82% of occurrence of nausea and vomiting. Post-operative nausea and vomiting occurred in 59% of the population that received greater than optimal prophylaxis. Researchers speculate that the high incidence of nausea and vomiting occurs due to potential damage of the vagal nerve during the operation. The motility of the stomach and intestines is also affected by the surgery and narcotics that patients take after the operation. Halliday and colleagues concluded that other methods of nausea and vomiting prevention should be evaluated in this population.

Aromatherapy and essential oils are an alternative method to controlling post-operative nausea and vomiting after post-surgical intervention. Although it has not been frequently studied in bariatric patients, it has been studied post-operatively for other surgeries and for vomiting after chemotherapy. According to a systematic review in 2012, three studies regarding post-operative nausea and vomiting found reduction in symptoms after inhalation of essential oils. The studies also noted reduction in need for nausea medication, improved patient satisfaction, and reduction in cost. A review by Cochrane and colleagues showed no reliable evidence of the effectiveness of peppermint oil. Other studies found that either peppermint or ginger were effective in the reduction of post-operative nausea and vomiting. However the studies had relatively small sample sizes and were not usually randomized control trials.

From the research and current studies, post-operative nausea and vomiting is a common complaint after bariatric surgery. Nausea relief inhalers could improve post-operative nausea and vomiting without the need for further medications, subsequently reducing the chance of side effects. This study could help improve patient satisfaction and increase the ability of the patient to ambulate after surgery with the use of a nausea relief inhaler.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old
* Attend the pre-operative class
* Must be able to read English
* Admitted to B4 surgical acute unit
* Surgery after May 31st, 2020

Exclusion Criteria:

* BMI greater than 60
* Pre-operatively on nausea medication
* Allergy to spearmint, lemon, ginger, and/or cedarwood
* History of Asthma or chronic obstructive pulmonary disease(COPD)
* Patient intubated or sedated for the 24 hours after surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-11-23 (Estimated); Study Completion 2024-11-23 (Estimated)

PRIMARY OUTCOMES:
Medication Administration Record | "Up to 24 hours"
  The amount of nausea and vomiting medication use will be determined by the medication administration record during chart review in the first 24 hours for each study patient.

SECONDARY OUTCOMES:
Rhodes index | "Up to 24 hours"
  Indicators of decreased stress and increased contentment will be found by patient's answers to questions regarding distress from dry heaving and retching and nausea and vomiting.
Length of stay | duration of hospital stay: date of discharge minus date of admittance)
  Length of stay will be tracked via chart review (date of discharge minus date of admittance)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Attaway, RN, Principal Investigator — Methodist Mansfield Medical Center
Locations (1):
- Methodist Mansfield Medical Center, Mansfield, Texas, United States

IPD SHARING:
Plan to Share IPD: No